CLINICAL TRIAL: NCT05181657
Title: LinkUP: COVID-19 Intervention for Underserved Populations Participating in Parent Study Proyecto La Frontera
Brief Title: LinkUP: COVID-19 Intervention for Underserved Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steffanie Strathdee, Distinguished Professor and Harold Simon Chair, Associate Dean of Global Health Sciences, Division of Infectious Disease and Global Public Health, UCSD Department of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LinkUP; R01DA049644 (NIH)
Record Dates: First submitted 2022-01-04; First posted 2022-01-06 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Motivational Interviewing
Keywords: Behavior change

STUDY DESIGN:
Intervention Model Description: The four OnPoint syringe exchange locations will be randomized to deliver either the active (intervention) or didactic (control) version of the LinkUP intervention. The randomization scheme will be developed using an algorithm by La Frontera's statistician. Half way into enrollment, there will be a one-week 'washout' period, after which time the two original intervention syringe exchange sites will become control sites and the two original control sites will become intervention sites. This cluster randomization scheme will help ensure that no neighborhood in San Diego County is denied access to the LinkUP intervention. By the end of the study, 75 LinkUP participants will have been randomized to an intervention site and 75 will have been randomized to a control site.
Who Masked: Participant, Investigator
Masking Description: Neither study participants or principal investigator will know which group participants have been assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LinkUP Active intervention (Experimental): The counselor will present basic evidence-based COVID-19 information on SARS-CoV-2 biology and epidemiology, testing and the safety and efficacy of available COVID-19 vaccines. The counselor will also address COVID-19 misinformation (e.g., that COVID is no worse than the flu), and COVID-19 disinformation (e.g., that COVID vaccines include a tracking device).
  The LinkUP active intervention combines education, motivational interviewing (MI), problem-solving, and ongoing support from peer counselors. Through an open discussion with one of OnPoint's peer counselors who are trained in MI, the counselor will present evidence-based COVID-19 information. Next, the counselor will attempt to identify the participant's concerns about COVID-19 and vaccination in an attempt to tip their decisional balance.
  Interventions: Behavioral: COVID-19 education
- LinkUP Control Condition (didactic intervention) (Placebo Comparator): As described above, the control condition is a one-way sharing of COVID-19 information presented by an OnPoint counselor. The counselor will be instructed to answer any questions the participant may have but will not engage in motivational interviewing counseling. The same educational materials used in the LinkUP intervention module will be used for this session and it will be completed within 45 minutes.
  Interventions: Behavioral: COVID-19 education

INTERVENTIONS:
Behavioral: COVID-19 education — This session will be completed within 45 minutes. The LinkUP intervention will be available in English and Spanish.

SUMMARY:
The goal of the present study is to evaluate a pilot intervention (LinkUP) to improve the uptake of COVID-19 testing and vaccination among PWID in San Diego County. Results will be shared with RADxUP consortium members, policymakers and program planners in California and across the US and used to estimate effect sizes for a future efficacy trial. Our study will inform efforts to leverage any of the 185 SSPs around the US as 'touchpoints' to reach marginalized communities, strengthening the nation's pandemic preparedness infrastructure to reduce COVID-19 health disparities.

DETAILED DESCRIPTION:
Together with our community partner, the Harm Reduction Coalition of San Diego's (HRCSD) OnPoint, a mobile safe syringe program (SSP), we will evaluate develop and evaluate an intervention to improve uptake of COVID-19 testing and vaccination. HRCSD's OnPoint will rely on UCSD's IRB review and approval for all aspects related to oversight of study and intervention implementation. Completion of primary endpoint data analyses was achieved on April 13, 2023. Study final completion date is January 31, 2024. Our Study Aims are :

1. To adapt an existing behavioral intervention incorporating motivational interviewing (MI) to improve uptake of HIV pre-exposure prophylaxis among people who inject drugs (PWID), by replacing the educational content with information intended to improve uptake of COVID19 testing and COVID19 vaccination.
2. To pilot test the intervention in Aim 1 (called LinkUP) at OnPoint's 4 mobile SSP locations across San Diego County. We expect that the LinkUP intervention will be acceptable to PWID and considered feasible and sustainable by OnPoint staff and the project's Community Scientific Advisory Board (CSAB).

ELIGIBILITY:
Inclusion Criteria

1. Enrolled in La Frontera,

   AND
2. Report NOT having been voluntarily tested for COVID-19 outside of La Frontera or report having had a mandatory COVID-19 test more than 2 months ago

   AND
3. a) Never vaccinated OR b) Received 1 shot of the Moderna vaccine (>=1 month ago) OR c) received 1 shot of the Pfizer vaccine (>=3 weeks ago) OR d) received 1 shot of the Jenssen vaccine (>=2 months ago) OR e) received 2 shots of the Moderna OR Pfizer vaccine (last shot >=5 months ago) OR f) received 1 shot of another vaccine (>=1 month ago) OR g) received 2 shots of another vaccine (last shot >=5 months ago). NOTE: participants who indicate that they were vaccinated but don't remember what vaccine they received would fall under the f category if they only received one shot and under the g category if they received 2 shots.

   OR
4. Enrolled in La Frontera AND report TWO or more of the following symptoms: a) new loss of smell or taste, b) cough, c) sore throat/congestion/runny nose, d) skin rash within the last week without having tested positive for COVID within the last month.

   OR
5. Enrolled in La Frontera AND report having EITHER fever/chills OR shortness of breath within the last week without having tested positive for COVID within the last month.

Exclusion Criteria

1. Not enrolled in La Frontera,

   AND
2. Report having been voluntarily tested for COVID-19 outside of La Frontera or report having had a mandatory COVID-19 test less than 2 months ago

   AND
3. a) Be vaccinated OR b) Received 1 shot of the Moderna vaccine (<1 month ago) OR c) received 1 shot of the Pfizer vaccine (<3 weeks ago) OR d) received 1 shot of the Jenssen vaccine (<2 months ago) OR e) received 2 shots of the Moderna OR Pfizer vaccine (last shot <5 months ago) OR f) received 1 shot of another vaccine (<1 month ago) OR g) received 2 shots of another vaccine (last shot <5 months ago). NOTE: participants who indicate that they were vaccinated but don't remember what vaccine they received would fall under the f category if they only received one shot and under the g category if they received 2 shots.

   OR
4. Not enrolled in La Frontera AND do NOT report TWO or more of the following symptoms: a) new loss of smell or taste, b) cough, c) sore throat/congestion/runny nose, d) skin rash within the last week without having tested positive for COVID within the last month.

   OR
5. Not enrolled in La Frontera AND do NOT report having EITHER fever/chills OR shortness of breath within the last week without having tested positive for COVID within the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steffanie Strathdee, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- La Frontera Project, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strathdee SA, Abramovitz D, Harvey-Vera AY, Stamos-Buesig T, Vera CF, Artamonova I, Logan J, Patterson TL, Servin AE, Bazzi AR. A Brief Peer-Led Intervention to Increase COVID-19 Vaccine Uptake Among People Who Inject Drugs in San Diego County: Results From a Pilot Randomized Controlled Trial. Open Forum Infect Dis. 2023 Jul 21;10(8):ofad392. doi: 10.1093/ofid/ofad392. eCollection 2023 Aug. PMID 37547856
- [Derived] Bazzi AR, Harvey-Vera A, Buesig-Stamos T, Abramovitz D, Vera CF, Artamonova I, Patterson TL, Strathdee SA. Study protocol for a pilot randomized controlled trial to increase COVID-19 testing and vaccination among people who inject drugs in San Diego County. Addict Sci Clin Pract. 2022 Sep 5;17(1):48. doi: 10.1186/s13722-022-00328-z. PMID 36064745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PWID, ≥18 years old, San Diego County residents who had not recently undergone voluntary COVID-19 testing were referred to mobile SSP sites. We randomized the 12 weeks of study implementation to involve either intervention or didactic-control condition administration (i.e., the study team administered the condition allocated to each particular week, regardless of SSP site). Counselors offered on-site rapid COVID-19 antigen testing. The LinkUP pilot RCT was conducted from March-June, 2022.
Units Other Than Participants: weeks
Groups:
- LinkUP Active Intervention: The counselor will present basic evidence-based COVID-19 information on SARS-CoV-2 biology and epidemiology, testing and the safety and efficacy of available COVID-19 vaccines. The counselor will also address COVID-19 misinformation (e.g., that COVID is no worse than the flu), and COVID-19 disinformation (e.g., that COVID vaccines include a tracking device).
  The LinkUP active intervention combines education, motivational interviewing (MI), problem-solving, and ongoing support from peer counselors. Through an open discussion with one of OnPoint's peer counselors who are trained in MI, the counselor will present evidence-based COVID-19 information. Next, the counselor will attempt to identify the participant's concerns about COVID-19 and vaccination in an attempt to tip their decisional balance.
  COVID-19 education: This session will be completed within 45 minutes. The LinkUP intervention will be available in English and Spanish.
Period: Overall Study
Arm/Group | LinkUP Active Intervention | LinkUP Control Condition (Didactic Intervention)
Started | 75; 5 weeks | 75; 7 weeks
Enrollment at the End of Week 1 | 0; 0 weeks | 7; 1 weeks
Enrollment at the End of Week 2 | 4; 1 weeks | 7; 1 weeks
Enrollment at the End of Week 3 | 4; 1 weeks | 11; 2 weeks
Enrollment at the End of Week 4 | 22; 2 weeks | 11; 2 weeks
Enrollment at the End of Week 5 | 22; 2 weeks | 23; 3 weeks
Enrollment at the End of Week 6 | 39; 3 weeks | 23; 3 weeks
Enrollment at the End of Week 7 | 39; 3 weeks | 39; 4 weeks
Enrollment at the End of Week 8 | 50; 4 weeks | 39; 4 weeks
Enrollment at the End of Week 9 | 50; 4 weeks | 60; 5 weeks
Enrollment at the End of Week 10 | 75; 5 weeks | 60; 5 weeks
Enrollment at the End of Week 11 | 75; 5 weeks | 72; 6 weeks
Enrollment at the End of Week 12 | 75; 5 weeks | 75; 7 weeks
Completed | 75; 5 weeks | 75; 7 weeks
Not Completed | 0; 0 weeks | 0; 0 weeks

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LinkUP Active Intervention | LinkUP Control Condition (Didactic Intervention) | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 38.0 [33.0 to 50.0] | 45.0 [36.0 to 54.0] | 40.5 [34.0 to 51.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 51 | 46 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 26 | 50
  Not Hispanic or Latino | 51 | 49 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 46 | 43 | 89
  More than one race | 18 | 20 | 38
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150
COVID-19 self-reported testing at baseline [Count of Participants; unit: Participants] | 33 | 34 | 67
On a scale of 1 to 10, how worried are you about getting COVID-19 (or getting it again)? [Median (Inter-Quartile Range); unit: units on a scale] — Question asked at baseline: On a scale of 1 to 10, how worried are you about getting COVID-19 (or getting it again)? NOTE: lower values mean less worry and higher values mean more worry.
  units on a scale | 5.0 [1.0 to 7.0] | 3.0 [1.0 to 6.0] | 4.0 [1.0 to 7.0]

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Testing
Description: Number of participants who agreed to and received onsite a COVID test right after receiving the intervention (i.e., same day as the intervention)
Time Frame: Day of the Intervention; The outcome for the last participant was ascertained on June 6th, 2022.
Measure: Count of Participants; unit: Participants
Arm/Group | LinkUP Active Intervention | LinkUP Control Condition (Didactic Intervention)
Number analyzed (Participants) | 75 | 75
Participants | 69 | 47
Statistical Analysis 1: Comparison: LinkUP Active Intervention vs LinkUP Control Condition (Didactic Intervention); To assess whether the active intervention was more successful than the control condition at increasing COVID-19 testing, we used univariable and multivariable Poisson regression models, with whether one received onsite testing right after the intervention as the outcome and intervention group as the main predictor. Potential clustering due to the randomization by week was accounted for by specifying an exchangeable correlation structure for participants who were recruited during the same week; Test type: Other — The intervention effect was determined via a two sided, 0.05 level of significance, multivariable Poisson regression model, with Intervention group as the primary predictor; p < 0.05, Poisson Regression — Alpha significance levels used: For the primary predictor (i.e., intervention group): alpha=0.05; For covariates: alpha=0.10; For interactions: alpha=0.15; Risk Ratio (RR) = 1.45, 95% CI 2-sided [1.18 to 1.78] — The estimate refers to the relative risk of getting a COVID-19 test onsite (Intervention/Control). Also, the above estimate is from the unadjusted Poisson regression model (i.e., model not adjusted for covariates and interactions)

2. Secondary Outcome: COVID-19 Vaccination
Description: Received ≥ one COVID shot within 6 months of intervention
  COVID-19 vaccination: Before trial started, SSP determined that limited staffing capacity to offer vaccination and addressing potential adverse events prevented this secondary outcome to be measured. Study participants were provided with referrals to community vaccine clinics throughout the County.
Time Frame: 6 months
Population: PWID in San Diego County who Participated in the Link-UP Intervention
Measure: Count of Participants; unit: Participants
Arm/Group | LinkUP Active Intervention | LinkUP Control Condition (Didactic Intervention)
Number analyzed (Participants) | 65 | 70
Participants | 15 | 12

ADVERSE EVENTS:
Time Frame: 6 months past baseline
Arm/Group | LinkUP Active Intervention | LinkUP Control Condition (Didactic Intervention)
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

LIMITATIONS AND CAVEATS:
1. Generalizability limited to study participants.
2. Recall, self-report of sensitive/socially stigmatized behaviors, COVID-19 measures not validated.
3. On-site COVID-19 vaccination not collected. Vaccination referrals provided instead.

Additional research to: a) confirm intervention efficacy and further explore the mechanisms of potential mediators and moderators of intervention effects and b) determine if LinkUP can effectively support COVID-19 vaccination uptake (our secondary outcome).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT05181657/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT05181657/ICF_001.pdf